CLINICAL TRIAL: NCT04208828
Title: IVIG for Drug and Device Refractory Gastrointestinal Auto-Immune Neuropathy
Acronym: GAIN
Status: Recruiting | Type: Observational
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Thomas Abell, Professor, University of Louisville
Other Study IDs: 15.0667
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Gastrointestinal Motility Disorder; Gastroparesis; Neuropathy
Keywords: Gastroparesis; Nausea; Vomiting; Abdominal Pain; Neuropathy
MeSH Terms: conditions — Gastroparesis; Nausea; Vomiting; Abdominal Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Patients with the symptoms of generalized GI dysmotility, including gastroparesis, are sometimes refractory to available medications, devices and other interventions/ Some of these patients have serologic and/or endo organ abnormalities and findings consistent with autoimmune neuropathies, primarily involving the GI tract. These disorders have been known as autoimmune gastrointestinal neuropathies (GAIN) or also as autoimmune gastrointestinal dysmotility (AGID), among other terms. Some patients respond to intravenous immunoglobulin (IVIG) and this study, which is an observational clinical series, documents the patients, their findings and standardized responses to therapy with IVIG.

DETAILED DESCRIPTION:
Gastrointestinal dysmotility disorders encompass a large group of patients including a subset with autoimmune findings, either on serologic testing and/or end organ anatomic and physiologic effects.

The identification of patients with autoimmune gastrointestinal neuropathies (GAIN) or also as autoimmune gastrointestinal dysmotility (AGID), has led to trial with autoimmune therapies. Most promising therapy has been intravenous immunoglobulin (IVIG) and this, usually given in 12-week courses with standard dosing, has helped a number of patient's refractory to other available therapies including diet, drugs, devices and enteral diversions/disruptions.This observational study documents clinical observations in consecutive patients meeting entry criteria who received IVIG.

Patients will have their gastrointestinal (GI) symptoms documented by a standardized patient reported outcome (PRO) survey at baseline and use the same assessment tools after at least one course of IVIG therapy.

ELIGIBILITY:
Inclusion Criteria: Patient with otherwise refractory symptoms of gastrointestinal (GI) motor disorders.

-

Exclusion Criteria: Inability to receive intravenous immunoglobulin.

-

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with GI motor disorders, including symptoms of gastroparesis, who are refractory to available dietary, drug, device, and endoscopic/surgical diversion therapies.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2028-01-02 (Estimated); Study Completion 2028-01-02 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal (GI) total symptoms score (TSS) | Baseline to latest, up to one year
  The primary outcome measures are patient symptoms via the traditional gastroparesis patient reported outcome scale. It uses a 0-4 scale from none to worse on GI Symptoms; for example: Nausea,Vomiting, Anorexia/Early Satiety, Bloating/distension, Abdominal Pain. Scored as each item plus a total that is the sum of the individual scales.The five Sx subscales of 0-4 each are summed for a total score range 0-20

CONTACTS AND LOCATIONS:
Locations (1):
- University of Louisville, Louisville, Kentucky, United States